CLINICAL TRIAL: NCT01550211
Title: Changes in Brain Synchronization During Perceptual and Linguistic Tasks in Schizophrenic Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shalvata Mental Health Center (Other)
Collaborators: Bar-Ilan University, Israel (Other)
Responsible Party: Sponsor
Other Study IDs: SHA-0001-12
Record Dates: First submitted 2012-03-07; First posted 2012-03-09 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Schizophrenic Patients

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Students: Healthy students from Bar-Ilan University
  Interventions: Device: Magnetoencephalograph (MEG)
- Schizophrenic patients' relatives: Healthy family members (parents or siblings) of the schizophrenic participants (chronic and naive)
  Interventions: Device: Magnetoencephalograph (MEG)
- Naive schizophrenic patients: Naive patients with a diagnosis of schizophrenia, a history of only one psychotic episode and un-medicated
  Interventions: Device: Magnetoencephalograph (MEG)
- Chronic schizophrenia patients: Chronic patients with a diagnosis of schizophrenia and a history of more than one psychotic episode
  Interventions: Device: Magnetoencephalograph (MEG)

INTERVENTIONS:
Device: Magnetoencephalograph (MEG) — Conducting a brain scan during a series of perceptual and linguistic tasks

SUMMARY:
This study aims to identify electrophysiological correlates of impaired perceptual and linguistic processes in chronic schizophrenic patients, un-medicated first-episode schizophrenic patients and their healthy relatives.

Following administrating some questionnaires (demographic details and psychiatric history questionnaire, handedness questionnaire, reading abilities test and positive and negative symptoms questionnaire) and performing a perception test and a verbal abstract intelligence test, participants will conduct a brain scan during a series of perceptual and linguistic tasks.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for chronic patients:

* Hebrew native speakers.
* Diagnosis of schizophrenia with a history of more than one episode.
* Capable and willing to provide informed consent.

Inclusion criteria for naive patients:

* Hebrew native speakers.
* Diagnosis of schizophrenia with a history of only one episode and unmedicated.
* Capable and willing to provide informed consent.

Inclusion criteria for patients' relatives (control group 1):

* Hebrew native speakers.
* Without any psychiatric history.
* Have a child and/or a sibling with schizophrenia.

Inclusion Criteria for students (control group 2):

* Hebrew native speakers.
* Without any psychiatric history.

Exclusion Criteria:

Exclusion Criteria for patient groups (chronic and "naïve"):

* Left handedness.
* Reading disability.
* Visual perception disability.
* Brain damage and/or a history of seizures.
* Impaired intelligence.
* Metal implants.

Exclusion Criteria for control groups (family members and students):

* Psychiatric history.
* Left handedness.
* Reading disability.
* Visual perception disability.
* Brain damage and/or a history of seizures.
* Impaired intelligence.
* Metal implants.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Chronic patients - Up to 30 chronic schizophrenic patients.
  2. Naive patients - Up to 30 unmedicated first episode schizophrenic patients.
  3. Patients' relatives - Up to 60 family members (parents or siblings) of the participants - control group 1.
  4. Students - Up to 30 students from Bar-Ilan University - control group 2.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2012-03; Primary Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Magnetic field amplitude and source | 45 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Hilik Levkovitz, Professor, Principal Investigator — Shalvata MHC
Locations (1):
- Shalvata MHC, Hod HaSharon, Israel